CLINICAL TRIAL: NCT03380650
Title: Study of Combined Use of Directional Atherectomy and Local Drug Delivery With Balloon Catheter System in the Treatment of Femoropopliteal Occlusive Disease
Brief Title: Study of DA+LDD in the Treatment of Femoropopliteal Occlusive Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-092
Record Dates: First submitted 2017-12-13; First posted 2017-12-21 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Peripheral Artery Disease; Endovascular Treatment
Keywords: femoropopliteal occlusive disease; directional atherectomy; local drug delivery; endovascular treatment
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: only the doctor know the group the patient goes into
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- durg-coated balloon dilation (Other): The drug-coated balloon will be used to treat the femoropopliteal occlusion.
  Interventions: Device: drug-coated balloon dilation
- directional atherectomy and LDD (Other): The directional atherectomy and local drug delivery will be used to treat the femoropopliteal occlusion.
  Interventions: Device: directional atherectomy and locol drug delivery

INTERVENTIONS:
Device: directional atherectomy and locol drug delivery — combined use of directional atherectomy and locol drug delivery for the treatment of femoralpopliteal disease
  Arms: directional atherectomy and LDD
Device: drug-coated balloon dilation — use of drug-coated balloon dilation for the treatment of femoralpopliteal disease
  Arms: durg-coated balloon dilation

SUMMARY:
This study will evaluate the effectiveness and safety of directional atherectomy plus local drug delivery using balloon catheter system in the treatment of femoropopliteal occlusive disease. Patients of femoropopliteal occlusive disease will randomly receive directional atherectomy plus local drug delivery using balloon catheter system and dilation using drug-coated balloon. Their clinical outcomes (e.g. 12-month late lumen loss rate, 1-year patency rate of target vessel) in 1 year after the treatment will be compared.

DETAILED DESCRIPTION:
Femoropopliteal occlusive disease is a common type of peripheral arterial disease. Endovascular treatment has been the first-line treatment of femoropopliteal occlusive disease. However, the in-stent re-stenosis has been a major limitation of well long-term patency rate after stent implantation. The chronic inflammation induced by stenting could be a main reason of re-stenosis. Then the concept "leave nothing behind" is proposed, and some novel treatment methods and devices, such as paclitaxel-coated balloon dilation, directional atherectomy, are developed. Directional atherectomy can effectively remove the atherosclerosis plaque but leave the inflammatory reaction along the atherectomy route. Here, we propose the hypothesis that using local drug delivery with balloon system can relieve the inflammation induced by atherectomy. Therefore, 40 patients of femoropopliteal occlusive disease will be randomly allocated into the group "directional atherectomy+local drug delivery with balloon system" or "drug-coated balloon only". The 1-year patency rate, incidence of complications, imaging parameters will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* age of 18-80 years old
* patients of femoropopliteal occlusive disease (Rutherford 2-4)
* length of lesion ≤ 20cm
* have signed the informed consent

Exclusion Criteria:

* serum Cr > 150 umol/L
* patients with acute thrombosis
* received endovascular treatment for femoropopliteal disease in recent 6 months
* less than 1 run-off vessel
* allergic to aspirin, heparin, clopidogrel, paclitaxel, contrast medium
* pregnancy and lactation
* relatively easy bleeding
* malignancy or irreversible organ failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
late lumen loss rate | 12 months
  the rate of late lumen loss of target vessel
patency rate | 6 months
  the rate of patency of target vessel
patency rate | 12 months
  the rate of patency of target vessel

SECONDARY OUTCOMES:
MLD | 12 months
  minimal lumen diameter of target vessel at 6 months
clinical outcomes | 12 months
  rate of re-intervention of target vessel
incidence of complications | 12 months
  incidence of treatment induced major complications
re-stenosis rate | 12 months
  the rate of re-stenosis (≥50)
adverse events | 12 months
  incidence of treatment related adverse events
Rutherford level | 12 months
  change of Rutherford level
ABI | 12 months
  change of ankle brachial index
main amputation | 12 months
  rate of main amputation

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhang, M.D., Ph.D., Principal Investigator — RenJi Hospital

IPD SHARING:
Plan to Share IPD: No